CLINICAL TRIAL: NCT02805270
Title: Implementation of a Medication Reconciliation Intervention and Its Impact on the Rate of ADEs and Healthcare Utilization 30 Days Following Discharge From the Hospital. A Randomized Controlled Trial.
Brief Title: Impact of Medication Reconciliation Intervention on the Rate of Preventable Adverse Drug Events (ADEs) and Healthcare Utilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MREC#715
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Adverse Drug Events
Keywords: adverse drug events, preventable, potential, counselling, medication reconciliation
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- medication reconciliation intervention (Experimental): medication reconciliation intervention comprises medication reconciliation on admission and discharge, bedside medication counseling and take-home medication list
  Interventions: Other: medication reconciliation intervention
- usual care (No Intervention): Usual care provided by ward pharmacist, nurses and doctors in the ward

INTERVENTIONS:
Other: medication reconciliation intervention — medication reconciliation intervention comprises medication reconciliation on admission and discharge, bedside medication counseling and take-home medication list
  Arms: medication reconciliation intervention

SUMMARY:
The implementation of a medication reconciliation intervention including: medication reconciliation on admission and discharge, bedside medication counselling and take-home medication list, on the development of adverse drug events within 30 days post discharge as primary outcome. Secondary outcome is the evaluation of its impact on health care resource utilization

DETAILED DESCRIPTION:
This is a randomized controlled trial in 587 patients randomized to intervention and usual care. The intervention is medication reconciliation on admission and discharge, bedside medication counselling and take-home medication list. Usual care is ward pharmacy practice. The primary outcomes are preventable and potential adverse drug events at 30 days post discharge. The secondary outcome is health care utilization: length of stay, emergency room visits, unplanned hospital visits, readmissions and travel abroad to seek medical attention.

ELIGIBILITY:
Inclusion Criteria:

* admitted to one of the two medical wards, male and female medical wards.
* was on at least one medication prior to admission
* spoke Arabic or English and can be (the patient or care giver) interviewed for medication history
* stayed in the hospital for at least 24 hours
* discharged on at least one chronic medication or is at least on one chronic medication even if not prescribed upon discharge

Exclusion Criteria:

* could not be interviewed due to language barrier, impaired cognition or other reasons and did not have a care giver
* was under specialties other than medical specialties, but was admitted to medical wards because of lack of beds in their respective wards
* was pregnant
* was already included in the study at a previous admission
* left the hospital against medical advice
* with length of stay of >60 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
number of patients with a preventable adverse drug event | 30 days
number of potential adverse drug events | 30 days

SECONDARY OUTCOMES:
number of emergency room visits | 30 days
number of unplanned hospital visits | 30 days
number of hospital readmissions | 30 days
number of patients who traveled abroad to seek second medical opinion | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Amna Al-Hashar, PhD candidate, Principal Investigator — Sultan Qaboos University College of Medicine and Health Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schnipper JL, Kirwin JL, Cotugno MC, Wahlstrom SA, Brown BA, Tarvin E, Kachalia A, Horng M, Roy CL, McKean SC, Bates DW. Role of pharmacist counseling in preventing adverse drug events after hospitalization. Arch Intern Med. 2006 Mar 13;166(5):565-71. doi: 10.1001/archinte.166.5.565. PMID 16534045
- [Background] Kripalani S, Roumie CL, Dalal AK, Cawthon C, Businger A, Eden SK, Shintani A, Sponsler KC, Harris LJ, Theobald C, Huang RL, Scheurer D, Hunt S, Jacobson TA, Rask KJ, Vaccarino V, Gandhi TK, Bates DW, Williams MV, Schnipper JL; PILL-CVD (Pharmacist Intervention for Low Literacy in Cardiovascular Disease) Study Group. Effect of a pharmacist intervention on clinically important medication errors after hospital discharge: a randomized trial. Ann Intern Med. 2012 Jul 3;157(1):1-10. doi: 10.7326/0003-4819-157-1-201207030-00003. PMID 22751755